CLINICAL TRIAL: NCT03627416
Title: A Pilot Study of Repetitive Transcranial Magnetic Stimulation for Improvement of Gait in Hereditary Spastic Paraplegia and Adrenomyeloneuropathy
Brief Title: Repetitive Transcranial Magnetic Stimulation as Therapy in Hereditary Spastic Paraplegia and Adrenomyeloneuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jakub Antczak (Other)
Responsible Party: Sponsor-Investigator, Jakub Antczak, Principal Investigator, Jagiellonian University
Organization: Jagiellonian University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: JagiellonianU59
Record Dates: First submitted 2017-10-23; First posted 2018-08-13 (Actual); Results first posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-08

CONDITIONS: Hereditary Spastic Paraplegia; Adrenomyeloneuropathy
Keywords: Hereditary spastic paraplegia; repetitive transcranial magnetic stimulation; disturbed gait; Adrenomyeloneuropthy
MeSH Terms: conditions — Spastic Paraplegia, Hereditary; Adrenoleukodystrophy

STUDY DESIGN:
Intervention Model Description: 16 patients with HSP or AMN will receive either active and sham stimulation in random order
Who Masked: Participant, Outcomes Assessor
Masking Description: Sham stimulation will be provided by holding the stimulating coil perpendicularly to the scalp, which assures similar impression as during active stimulation but prevents significant magnetic field to reach the brain tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active rTMS (Experimental): 10 hertz (Hz) rTMS will be administered over bilateral primary motor areas for the muscles of lower extremities. Therapy will include five daily sessions (on consecutive week days). In every sessions 3000 magnetic pulses of 90% of the resting motor threshold intensity will be elicited.
  Interventions: Device: rTMS
- Sham rTMS (Sham Comparator): Sham stimulation will mimic the active one except that the stimulating coil will be held perpendicularly to the scalp, which assures similar impression as the active stimulation but prevents that significant magnetic field will reach brain tissue.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — high frequency rTMS to induce the long term potentiation of primary motor areas for the muscles of lower extremities

SUMMARY:
Hereditary spastic paraplegia (HSP) is the group of inherited disorders, characterized by progressive gait disturbance. There is no established therapy. Adrenoleukodystrophy (AMN) is an x-linked hereditary disease. One of its form, the adrenomyeloneuropathy has the same symptoms as HSP. Current therapeutic options for AMN are very limited. Repetitive Transcranial Magnetic Stimulation (rTMS) is a noninvasive method of modulation of brain plasticity. The purpose of this study is to compare the effectiveness of rTMS in improving the HSP- and AMN-related gait disturbance and other symptoms with sham stimulation.

Intervention will include five daily sessions. In each session 1500 magnetic pulses will be administered to each of both primary motor areas for lower extremities. Assessment of gait and of strength and spasticity of lower extremities will be made before and after therapy, as well as two weeks later.

DETAILED DESCRIPTION:
Hereditary spastic paraplegia (HSP) is a group of inherited disorders, characterized by progressive gait disturbance with weakness and spasticity, which predominate in lower extremities. There is no established therapy. Adrenoleukodystrophy (AMN) is an x-linked hereditary disease. One of its form, the adrenomyeloneuropathy has the same symptoms as HSP. Current therapeutic options for AMN are very limited. Repetitive Transcranial Magnetic Stimulation (rTMS), a noninvasive method of modulation of brain plasticity proved to be effective in improving the gait performance in several conditions such as Parkinson Disease, vascular Parkinsonism, partial spinal cord injury and in post-stroke paresis. Previous studies documented also altered cortical excitability in HSP patients.

The purpose of this study is to compare the effectiveness of 10 hertz (Hz) rTMS over the primary motor cortices in improving the gait and strength and spasticity of lower extremities with sham stimulation in HSP and AMN patients.

Intervention will include five daily sessions. In each session 1500 magnetic pulses will be administered to each of both primary motor areas for lower extremities. Assessment of gait and of strength and spasticity of lower extremities will be made before and after therapy, as well as two weeks later.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of hereditary spastic paraplegia - confirmed genetically, on the basis of family history or on exclusion or diagnosis of adrenomyeloneuropathy - confirmed genetically or by the elevated plasma very long chain fatty acid or on family history
* Gait disturbances affecting daily activities
* Ability to walk 10 meters without assistance or with crutches or with rollator walker

Exclusion Criteria:

* Presence of signs or symptoms indicating other than HSP or AMN ethiology of gait disturbances
* Contraindications for rTMS as listed by the Guidelines of the International Federation of Clinical Neurophysiology (IFCN 2009) i.e. seizure in the past, epilepsy, presence of magnetic material in the reach of magnetic field, pregnancy, likelihood to get pregnant, intracranial electrodes, cardiac pacemaker or intracardiac lines, frequent syncopes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jakub M Antczak, MD, Principal Investigator — Jagiellonian University Medical College, Department of Neurology
Locations (1):
- Jagiellonian University Medical College, Department of Neurology, Krakow, Poland

REFERENCES:
- [Result] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Derived] Antczak J, Pera J, Dabros M, Kozminski W, Czyzycki M, Wezyk K, Dwojak M, Banach M, Slowik A. The Effect of Repetitive Transcranial Magnetic Stimulation on Motor Symptoms in Hereditary Spastic Paraplegia. Neural Plast. 2019 May 12;2019:7638675. doi: 10.1155/2019/7638675. eCollection 2019. PMID 31214256

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 15 patients meeting inclusion criteria. One patient dropped out due to seizure, when he was in active treatment.
Groups:
- Active rTMS First, Then Sham rTMS: First intervention: 10 hertz (Hz) rTMS will be administered over bilateral primary motor areas for the muscles of lower extremities. Therapy will include five daily sessions (on consecutive week days). In every sessions 3000 magnetic pulses of 90% of the resting motor threshold intensity will be elicited.
  The washout will last at least one month.
  Second intervention:
  Sham stimulation will mimic the active one except that the stimulating coil will be held perpendicularly to the scalp, which assures similar impression as the active stimulation but prevents that significant magnetic field will reach brain tissue.
  rTMS: high frequency rTMS to induce the long term potentiation of primary motor areas for the muscles of lower extremities
- Sham rTMS, Then Active rTMS: First intervention: Sham stimulation will mimic the active one except that the stimulating coil will be held perpendicularly to the scalp, which assures similar impression as the active stimulation but prevents that significant magnetic field will reach brain tissue.
  The washout will last at least one month.
  Second intervention: 10 hertz (Hz) rTMS will be administered over bilateral primary motor areas for the muscles of lower extremities. Therapy will include five daily sessions (on consecutive week days). In every sessions 3000 magnetic pulses of 90% of the resting motor threshold intensity will be elicited.
  rTMS: high frequency rTMS to induce the long term potentiation of primary motor areas for the muscles of lower extremities
Period: Overall Study
Arm/Group | Active rTMS First, Then Sham rTMS | Sham rTMS, Then Active rTMS
Started | 8 | 7
Completed | 8 | 6
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Active rTMS, Then Sham rTMS: First intervention:
  10 hertz (Hz) rTMS will be administered over bilateral primary motor areas for the muscles of lower extremities. Therapy will include five daily sessions (on consecutive week days). In every sessions 3000 magnetic pulses of 90% of the resting motor threshold intensity will be elicited.
  The washout period will last at least one month.
  Second intervention:
  Sham stimulation will mimic the active one except that the stimulating coil will be held perpendicularly to the scalp, which assures similar impression as the active stimulation but prevents that significant magnetic field will reach brain tissue.
  rTMS: high frequency rTMS to induce the long term potentiation of primary motor areas for the muscles of lower extremities
- Sham rTMS, Then Active rTMS: First intervention:
  Sham stimulation will mimic the active one except that the stimulating coil will be held perpendicularly to the scalp, which assures similar impression as the active stimulation but prevents that significant magnetic field will reach brain tissue.
  The washout period will last at least one month.
  Second intervention:
  10 hertz (Hz) rTMS will be administered over bilateral primary motor areas for the muscles of lower extremities. Therapy will include five daily sessions (on consecutive week days). In every sessions 3000 magnetic pulses of 90% of the resting motor threshold intensity will be elicited.
  rTMS: high frequency rTMS to induce the long term potentiation of primary motor areas for the muscles of lower extremities
- Total: Total of all reporting groups
Arm/Group | Active rTMS, Then Sham rTMS | Sham rTMS, Then Active rTMS | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (11.9) | 41.7 (7.5) | 44.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 6 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Poland | 8 | 7 | 15
Central motor conduction time [Mean (Standard Deviation); unit: milliseconds] | 18.2 (3.4) | 20.3 (6.6) | 19.1 (5.2)
Amplitude of motor evoked potentials [Mean (Standard Deviation); unit: millivolts] | 1.1 (0.6) | 0.7 (0.5) | 0.9 (0.5)
Motor threshold for left abductor hallucis [Mean (Standard Deviation); unit: percentage of the maximal stimulator out] | 64.1 (7.5) | 63.5 (8.0) | 63.9 (7.7)
Motor threshold for the right abductor hallucis [Mean (Standard Deviation); unit: Percentage of the max stimulator output] | 61.4 (12.1) | 62.8 (8.3) | 62.0 (10.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Walking Time in 10 Meter Walk Test to the Measurement Taken Directly After rTMS
Description: Change in time of walking barefoot the distance of 10 meters with maximal speed, but safely, between baseline and directly after rTMS.
Time Frame: Before rTMS, directly (on the same day) after rTMS
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 14 | 14
seconds | -5.41 (16.42) | 1.70 (8.52)

2. Secondary Outcome: Change in Timed up and go Test
Description: Time of standing up from a chair, walking three metres to cross a line drawn 3 meters ahead and going back to sit down on the chair.
Time Frame: Baseline, directly (on the same day) after rTMS and 14 days later
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 14 | 14
seconds
  Baseline vs. after rTMS | -4.72 (13.90) | 0.18 (4.83)
  Baseline vs. 14 days later | -2.92 (7.29) | 0.78 (7.24)

3. Secondary Outcome: Change in Medical Research Council Scale (MRC)
Description: Change in bilateral assessment of the strength of following movements: hip flexion, knee flexion and extension, ankle flexion and extension. Assessment will be made according to six degrees (0 to 5) MRC scale, with higher values representing stronger movements, which is better outcome. Values are averaged from all movements tested.
Time Frame: Baseline, directly (on the same day) after rTMS and 14 days later
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 14 | 14
score on a scale
  Baseline vs. directly after rTMS | 0 (0) | 0.06 (0.22)
  Baseline vs. 14 days later | 0.09 (0.27) | 0 (0.32)

4. Secondary Outcome: Modified Ashworth Scale
Description: Bilateral assessment of spasticity in following movements: hip flexion, knee flexion and extension, ankle flexion and extension. Assessment will be made according to six degrees (0 to 5) Modified Ashworth Scale, with higher values representing more severe spasticity, which is worse outcome. Values are averaged from all movements tested.
Time Frame: Baseline, directly (on the same day) after rTMS and 14 days later
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 14 | 14
score on a scale
  Baseline vs. after rTMS | -0.36 (0.50) | 0 (0.46)
  Baseline vs. 14 days later | -0.27 (0.46) | -0.11 (0.53)

5. Secondary Outcome: Change From Baseline Walking Time in 10 Meter Walk Test to the Measurement Taken Two Weeks After rTMS
Description: Change in time of walking barefoot the distance of 10 meters with maximal speed, but safely, between baseline and 14 days after finishing rTMS therapy.
Time Frame: Baseline, 14 days after rTMS
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 14 | 14
seconds | -5.84 (17.52) | 0.93 (6.54)

ADVERSE EVENTS:
Time Frame: 2 years.
Arm/Group | Active rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15
Other Adverse Events (participants affected / at risk) | 4/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS (N=15) | Sham rTMS (N=15)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) — In one patient a seizure occurred during the third session of real stimulation. It began with a tonic flexion of the hip and knee. Then, a loss of consciousness and generalized convulsions followed. The seizure resolved after three minutes.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS (N=15) | Sham rTMS (N=15)
Sleplessness (Nervous system disorders) | 1 (1) | 0 (0) — One female participant (62 years of age) complained about sleeplessness after the first two sessions of active stimulation.
Head ache (Nervous system disorders) | 3 (3) | 0 (0) — Mild head ache during first sessions of active rTMS

LIMITATIONS AND CAVEATS:
Limited number of sessions, which may decrease the magnitude of the therapeutic effect.

The abundant pharmacotherapy with baclofen could considerably reduce observed effects on spasticity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT03627416/Prot_SAP_000.pdf